CLINICAL TRIAL: NCT00868712
Title: Warfarin and Coronary Calcification Project
Acronym: WACC
Status: Completed | Type: Observational
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Todd C. Villines, Director, Cardiovascular Research, Walter Reed Army Medical Center
Other Study IDs: WU# 04-12020
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Results first posted 2012-08-24 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Coronary Calcification
Keywords: coronary calcification; vitamin K dependent proteins; warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Warfarin use < 6 months
- 2: Warfarin use 6-24 months
- 3: Warfarin use >24 months

SUMMARY:
The purpose of the study is to assess whether the use of warfarin, a commonly used anticoagulation drug, is associated with increased amounts of coronary artery calcification. Studies in animals and preliminary but small retrospective studies in humans have suggested a possible link to increased tissue calcification with use of this drug. The researchers will investigate this by assessing the amount of calcification seen in the coronary arteries using a specialized computed tomography (CT) scan (electron-beam CT) and assessing to see if the amount is influenced by the amount of time a patient has been taking warfarin. The researchers will exclude patients with known coronary artery disease, chronic kidney disease or hyperparathyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older
* Patients referred to begin or already treated with warfarin anticoagulation therapy.

Exclusion Criteria:

* Known prior myocardial infarction or coronary heart disease
* History of advanced chronic kidney disease manifested by serum creatinine>2 or calculated glomerular filtration rate (GFR)<30
* History of hyperparathyroidism
* Current hypercalcemia
* Current hyperphosphatemia
* Uncertain duration of warfarin therapy
* Lack of records documenting international normalized ratio (INR) during therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients without known coronary heart disease, disorders of calcium metabolism or chronic kidney disease aged > 18 years who are referred to take or currently taking warfarin and are followed in the Anticoagulation Management Clinic at Walter Reed Army Medical Center (WRAMC).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2004-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Villines TC, O'Malley PG, Feuerstein IM, Thomas S, Taylor AJ. Does prolonged warfarin exposure potentiate coronary calcification in humans? Results of the warfarin and coronary calcification study. Calcif Tissue Int. 2009 Dec;85(6):494-500. doi: 10.1007/s00223-009-9300-4. Epub 2009 Oct 22. PMID 19847375
- See also: Publication abstract — http://www.ncbi.nlm.nih.gov/pubmed/19847375

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment is complete. All patients were recruited from within the Walter Reed Anticoagulation Clinic, as specified in the protocol.
Groups:
- Warfarin Use Short Duration: Warfarin use for less than 6 months
- 2 - Warfarin Use Intermediate: Warfarin use for 6 to 24 months in duration
- 3 - Warfarin Use Chronic: Warfarin use >24 months
Period: Overall Study
Arm/Group | Warfarin Use Short Duration | 2 - Warfarin Use Intermediate | 3 - Warfarin Use Chronic
Started | 31 | 11 | 28
Completed | 31 | 11 | 28
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Warfarin Use Short Duration | 2 - Warfarin Use Intermediate | 3 - Warfarin Use Chronic | Total
Number analyzed (Participants) | 31 | 11 | 28 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 4 | 9 | 34
  >=65 years | 10 | 7 | 19 | 36
Age Continuous [Mean (Standard Deviation); unit: years] | 64 (13) | 68 (11) | 73 (12) | 68 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 9 | 24
  Male | 21 | 6 | 19 | 46
Region of Enrollment [Number; unit: participants]
  United States | 31 | 11 | 28 | 70

OUTCOME MEASURES:

1. Primary Outcome: Coronary Calcification (Presence and Degree as Measured by Agatston Score) Attributed to Duration of Warfarin Use in Months After Controlling for Standard Cardiovascular Risk Factors to Include the Framingham Risk Score
Description: The Agatston score is calculated using a non-contrast computed tomography (CT) scan to measure for the presence and severity of coronary artery disease through identification of calcification in the coronary arteries. Scores can range from 0 to several thousands. The measure is without units. Score categories are as follows: 0 = no coronary disease; 1-100 = low amount of coronary artery disease; 101-400 = moderately elevated score / moderate coronary artery disease; 401-1000 = severely elevated score; >1000 very severely elevated score. Higher Agatston scores corelate with more coronary artery disease and predict a higher risk of coronary heart disease events and mortality.
Time Frame: EBCT scan is done at time of enrollment of patient into 1 of 3 groups based on warfarin use duration: <6 months; 6-24 months; >24 mos.
Population: After interim analysis following n=70 showed no effect, further enrollment was halted.
Measure: Mean (Standard Deviation); unit: Agatston Score
Arm/Group | Warfarin Use Short Duration | 2 - Warfarin Use Intermediate | 3 - Warfarin Use Chronic
Number analyzed (Participants) | 31 | 11 | 28
Agatston Score | 175 (285) | 289 (382) | 426 (789)

2. Secondary Outcome: International Normalized Ratio
Description: The International Normalized Ratio (INR) is a standardized lab value that measures the intensity of anticogulation using warfarin. It is used to monitor patients taking warfarin.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Warfarin Use Short Duration | 2 - Warfarin Use Intermediate | 3 - Warfarin Use Chronic
Number analyzed (Participants) | 31 | 11 | 28
ratio | 1.8 (0.9) | 2.4 (0.4) | 2.5 (0.4)

ADVERSE EVENTS:
Time Frame: 1 month (until calcium scan completed).
Arm/Group | Warfarin Use Short Duration | 2 - Warfarin Use Intermediate | 3 - Warfarin Use Chronic
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/11 | 0/28
Other Adverse Events (participants affected / at risk) | 0/31 | 0/11 | 0/28

LIMITATIONS AND CAVEATS:
Cross-sectional nature, small sample size. Initially powered for sample size of 100 subjects, our trial was stopped early after an interim analysis at 70 subjects demonstrated no trend for effect of warfarin after adjusting for standard risk factors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes